CLINICAL TRIAL: NCT05940311
Title: Versatile Ampification Method for Single-Molecule Detection in Liquid Biopsy
Brief Title: Versatile Ampification Single-Molecule Detection in Liquid Biopsy
Acronym: VerSiLiB
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: VTT Technical Research Centre, Finland (Other); Institute of Health Information and Statistics of the Czech Republic (Other Government); Universita degli Studi di Catania (Other); FINNADVANCE (FIN) (Unknown); PDC Biotech GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RS1685/22 (2670)
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Liquid Biopsy; Melanoma (Skin); Melanoma Stage III; Melanoma Stage IV
Keywords: BRAFV600E
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection; Circulating Tumor DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood drowing in K2EDTA vacutainer to obtain plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood sampling in addition to the blood normally required for their clinical management — Patients will undergo blood sampling in addition to the blood normally required for their clinical management. The study aims to collect 50 blood samples (one to 4) from 20 patients undergoing treatment in the adjuvant or advanced (metastatic) setting, as per standard of care. The first blood sample (T1) will be carried out immediately before the treatment, the subsequent blood samples (T2-T4) will coincide with the periodic radiographic re-evaluations, typically at months 3 and 6 (M3 and M6, T2 and T3), and at progression/recurrence, if and when recorded.
Procedure: Blood plasma and circulating tumor DNA (ctDNA) — Blood drawing by venepuncture (elbow) in K2EDTA vacutainers to obtain blood plasma.The patients will otherwise receive the most appropriate treatment for their condition. The following data will be collected and pseudo-anonymised: demographic data (age and gender), histopathology including primary and metastatic sites, BRAF status, medical imaging, previous therapies assigned if any

SUMMARY:
The trial will test a paradigm-changing in vitro diagnostic device for Liquid Biopsy enabling facile simultaneous detection of protein and nucleic acid analytes with sensitivity at single-molecule level, e.g. not achievable with any alternative technology. A novel affinity-mediated transport amplification (AMT) method will be tested allowing for the multiplexed quantification of rare biomarkers circulating in blood. The Versilib AMT photonic biosensor will test two analytes: the known actionable DNA mutation BRAF p.V600E, and a melanoma-restricted protein antigen. The results will be compared to digital PCR and ELISA methods.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥ 18
* PFS≤2
* Patients willing to sign an informed consent;
* Confirmed (cytologically or histologically) cutaneous melanoma diagnosis
* Confirmed BRAF p. V600E tumor status
* Eligible for BRAFi/MEKi treatment or Immune checkpoint blockade in either the adjuvant or advanced settings (the latter typically stages III/IV, high risk).

Exclusion Criteria:

* Life expectancy <8 weeks
* Other clinical conditions preventing blood drawing compliance, as per physician's choice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BRAF V600E Melanoma patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pilot study, descriptive statistics will be adopted (frequency, average, standard deviation, median, interval). Concordance indexes will be calculated, e.g. between dPCR and ELISA assays on the one hand and Versilib data on the other. | 48 months
  Concordance will determine whether the Versilib approach is technically feasible, e.g. whether method is sound, tests meet minimal requirements (technical sensitivity, reproducibility, accuracy). False positives and false negatives will be assessed. The results of descriptive statistics will be the basis to elaborate specific hypotheses (e.g. clinical scenarios) that will be the subject of future studies.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.versilib.eu